CLINICAL TRIAL: NCT03264300
Title: Development and Validation of Advanced MRI Methods for Clinical Applications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Arnold, Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHXA-16-0235-10-08; 1R01CA213158-01A1 (NIH)
Record Dates: First submitted 2017-07-11; First posted 2017-08-29 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumor
Keywords: brain tumor, MRI
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Development of advanced MRI methods (Active Comparator): Subjects with brain tumor. Subjects may be scanned using a single time-point to permit development and optimization of advanced MRI methods. Subjects may be scanned up to two times, with both visits occurring within one month, to permit analysis of test-retest reliability/repeatability.
  Interventions: Other: MRI
- Validation of rCBV accuracy (Active Comparator): 64 subjects with primary glioma and 96 subjects with recurrent glioma. Subjects will be scanned using a single time-point to validate rCBV accuracy.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI scans to include: scout images, transmitter tuning, shimming, slice prescription - 5 min; conventional structural MRI; T1-weighted anatomic MRI scan - 7 min; and, T2-weighted anatomic MRI scan - 5 min. Advanced MRI to include: Diffusion Weighted MRI (DW-MRI) - 7 min; Chemical Exchange Saturation Transfer (CEST) - 9 min; Dynamic Susceptibility Contrast / Dynamic Contrast Enhanced MRI - 8 min; and, other advanced imaging, as needed, to be determined. Post-contrast conventional MRI to include T1-weighted anatomic MRI scan - 7 min. Repeat within 1 month.
  Arms: Development of advanced MRI methods
Other: MRI — MRI scans to include: scout images, transmitter tuning, shimming, slice prescription - 5 min. Conventional structural MRI to include: T1-weighted anatomic MRI scan - 7 min; and, T2-weighted anatomic MRI scan - 5 min. Serial DSC-MRI: staged injections of Gd-based contrast and Ferumoxytol - 20 min. Post-contrast conventional MRI: T1-weighted anatomic MRI scan - 7 min.
  Arms: Validation of rCBV accuracy

SUMMARY:
A critical aspect of brain tumor patient management is the radiographic assessment of tumor status, which is used for diagnosis, localization, surgical planning and surveillance. The primary goal is to develop and apply advanced, quantitative magnetic resonance imaging (MRI) techniques that can supplement existing high-resolution anatomic imaging to aid clinical decision-making for patients diagnosed with brain tumors. The studies proposed herein involve the development of advanced imaging methods that are intrinsically sensitive to the biophysical characteristics associated with tumor pathogenesis, as they are more likely to improve tumor characterization and localization and may offer early and more specific indicators of treatment response. These advanced methods include diffusion-weighted imaging (DWI), chemical exchange saturation transfer (CEST), and dynamic susceptibility contrast (DSC) perfusion MRI. A secondary objective of this study is to validate cerebral blood volume (CBV) metrics acquired using a DSC acquisition and post-processing methods by comparison with an intravascular reference standard contrast agent. Validated perfusion imaging techniques will improve the reliability and relevancy of derived CBV metrics across a range of clinical applications, including tumor localization, treatment guidance, therapy response assessment, surgical and biopsy guidance, and multi-site clinical trials of conventional and targeted brain tumor therapies.

DETAILED DESCRIPTION:
The objectives of this study are to (1) Develop and optimize acquisition methods for MRI-based biomarkers that are indicative of brain tumor pathophysiology. These methods include, but are not limited to, DWI, CEST, and Dynamic Susceptibility Contrast (DSC) and Dynamic Contrast Enhanced (DCE) MRI; and (2) Validate DSC-MRI accuracy by comparison to an intravascular reference standard. Developmental studies: During the development of new imaging-based biomarkers, it is critical to optimize acquisition parameters, systematically characterize performance and contrast in the pathology of interest, validate with histopathology and establish test-retest repeatability. Thus, the first goal of this study is to develop advanced Diffusion Weighted Imaging (DWI), CEST and DSC/DCE-MRI methods for application to brain tumors. Objective 1 is a single-center study of up to 60 subjects being done to explore and optimize imaging signatures indicative of altered functional tumor states. These advanced imaging methods will allow the investigators to probe neuropathological tumor correlates, including cellular characteristics, molecular and metabolic changes, and vascular characteristics. Compared to existing conventional anatomic imaging, the researchers hypothesize that these experimental methods will be better able to characterize brain tumors and will have the potential to serve as new biomarkers of diagnostic and therapeutic importance. The researchers approach brings together biophysical and physiological information obtained from MRI and correlates this with clinical diagnoses and outcomes. Validation of DSC-MRI: Despite DSC-MRI's potential impact on clinical care, its broad scale integration has been slow, in large part from a lack of consensus about methodology and how to prevent potential CBV inaccuracies. Although DSC-MRI relies on the assumption that gadolinium-based contrast agents remain within the vascular lumen, this condition is often violated in vivo. If not corrected for, contrast agent leakage effects lead to CBV inaccuracy, misdiagnosis, and potentially mistreatment. While there exist numerous leakage correction strategies that have been shown to clearly improve DSC-MRI's clinical utility (e.g., predicting therapeutic response), a key limitation has prevented the standardization and wide-spread adoption of DSC-MRI methodology: To date, no study has validated the accuracy of leakage corrected CBV measures in patients. So while leakage corrected CBV values may be used, for example, to differentiate tumor recurrence from post-treatment effects, it is unknown whether this clinical benefit is a consequence of the complex combination of pulse sequence parameters, kinetics, dosing scheme, relaxivities, and leakage correction strategy or if the computed CBV actually reflects the underlying vascular density. This distinction is critical because it has implications for DSC-MRI standardization, establishing CBV thresholds for clinic use, multi-site comparisons and clinical trials. The investigators believe this limitation represents the most critical and clinically relevant challenge in the field of brain tumor DSC-MRI that urgently needs to be addressed. Objective 2 is a single-center study of up to 160 subjects being done to validate the accuracy of DSC-MRI measures of CBV. To validate the DSC-MRI measures derived from small molecular weight gadolinium-based (Gd) contrast agents, the investigators will compare rCBV maps to those derived from the intravascular contrast agent, Ferumoxytol. Ferumoxytol has been evaluated in humans as a potential DSC-MRI contrast agent but not for the purposes of validating leakage correction techniques. Since ferumoxytol-based DSC-MRI is not influenced by leakage effects, it enables the assessment of the most reliable perfusion metrics that can be expected from DSC-MRI and, as such, is the most reliable reference standard by which to evaluate CBV accuracy. Note that while ferumoxytol is undergoing clinical trials as a potential DSC-MRI contrast agent, it is unlikely to replace Gd-based contrast agents because it cannot provide the signal enhancement expected on conventional post-contrast T1-weighted images and is therefore unsuitable for use with standard response criteria.

ELIGIBILITY:
Inclusion Criteria:

* Must have either radiological or established histological diagnosis of the following: glioma / central nervous system (CNS) lymphoma / meningioma or brain metastases.
* Willing and able to provide written informed consent in compliance with the regulatory requirements. If a subject is unable to provide written informed consent, written informed consent may be obtained from the subject's legal representative.
* In the opinion of the investigator, able to fully participate in the study and sufficiently proficient in English to be capable of reliably completing study assessments.
* Sexually active women of child-bearing potential (Groups 1 and 2) and men (Group 2 only) must agree to use adequate methods to avoid pregnancy.

Exclusion Criteria:

* Subjects who have a contraindication for MRI: presence of an incompatible bio-implants (e.g., pacemakers, neurostimulators, electronic infusion pumps, etc.), metal in their bodies (non-MRI compatible cerebral aneurysm clips, shrapnel, metallic fragments in or near the eyes as pertains to metal workers and machinists), or noticeable anxiety and/or claustrophobia and/or severe vertigo when moved into the magnet bore.
* Subjects who are pregnant or lactating or who suspect they might be pregnant.
* (Groups 1 and 2, subjects receiving intravenous gadolinium (Gd) contrast material). Subjects with renal insufficiency or known allergy to Gd-based contrast material.
* (Group 2 only) Subjects with known or suspected iron overload.
* (Group 2 only) Subjects with known allergic or hypersensitivity reactions to parenteral iron treatment or other intravenous iron products; subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion.
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
* Any other reasons that, in the opinion of the Investigator, the candidate is determined to be unsuitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2022-06-26 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
cerebral blood volume | Within 60 days of MRI
  In patients with brain tumors we will develop and optimize advanced MRI methods to characterize blood volume.
the contrast agent extravasation rate constant (Ktrans, 1/min) | Within 60 days of MRI
  In patients with brain tumors we will develop and optimize advanced MRI methods to characterize Ktrans
Repeatability coefficient | within 60 days of MRI
  will assess the repeatability of MRI

SECONDARY OUTCOMES:
Intraclass correlation coefficient | Within 60 days of MRI
  Validate DSC-MRI accuracy by comparison to an intravascular reference standard by comparing rCBV maps to those derived from the intravascular contrast agent, Ferumoxytol

CONTACTS AND LOCATIONS:
Overall Officials: C C Quarles, PhD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix; Ashley M Stokes, PhD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States